CLINICAL TRIAL: NCT03804164
Title: A Study of the Feasibility and Acceptability of a Psycho-Educational Cognition Intervention in Adolescents and Young Adults (AYAs) With Cancer
Brief Title: Psycho-Educational Cognition Intervention in Patients With Blood and Lymph Cancer
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Feasibility
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 18442; NCI-2018-03851 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 18442 (Other: City of Hope Medical Center)
Record Dates: First submitted 2019-01-11; First posted 2019-01-15 (Actual); Last update posted 2020-12-17 (Actual); Status verified 2020-12

CONDITIONS: Hematopoietic and Lymphoid Cell Neoplasm
MeSH Terms: conditions — Hematologic Neoplasms | interventions — Early Intervention, Educational; Educational Status; Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Supportive Care (psycho-educational sessions) (Experimental): Patients participate in a psycho-educational program weekly over 2 hours for 6 weeks.
  Interventions: Other: Educational Intervention; Other: Quality-of-Life Assessment; Other: Survey Administration

INTERVENTIONS:
Other: Educational Intervention — Attend Emerging from the Haze psychoeducational sessions
  Other Names: Education for Intervention; Intervention by Education; Intervention through Education; Intervention, Educational
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Survey Administration — Ancillary studies

SUMMARY:
This pilot trial studies how well a psycho-educational program called Emerging from the Haze works in helping patients with blood and lymph cancer. Sometimes, patients who have undergone treatment for cancer experience thinking or memory problems that make work, school, or everyday life activities, such as grocery shopping, difficult. The Emerging from the Haze program may provide resources to help deal with these types of challenges in patients with blood and lymph cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Demonstrate feasibility and acceptability for young adult survivors of various cancers utilizing Emerging from the Haze program.

SECONDARY OBJECTIVES:

I. Describe, summarize study population. II. Characterize, compare the measure scores at pre-intervention assessment to the measure scores at post-intervention assessment.

OUTLINE:

Patients participate in the Emerging from the Haze psycho-educational program weekly over 2 hours for 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of a hematological malignancy.
* Having received chemotherapy with or without radiation therapy.
* Physician approval.
* Functional Assessment of Cancer Therapy-Cognition (FACT-COG) score < 59 on the perceived cognitive impairments (PCI) subscale.
* Eligible after 2 months (60 +/- 5 days) of completing all their active cancer treatment with the exception of patients that are post-transplant.
* Subjective complaint of cognitive concerns at time of enrollment.
* Must be able to understand and communicate proficiently in English.
* Ability to understand and the willingness to sign a written informed consent.
* Agree to complete study surveys.

Exclusion Criteria:

* Patients who have significant personality disorders or unstable psychiatric disorders as assessed by the interviewing clinician.
* Patients with known brain metastases, history of brain metastases or radiation to the brain.
* Patients with a history of stroke or other pre-existing neurological condition that may contribute to cognitive dysfunction.
* Non-English speaking patients.

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2020-02-10 (Actual); Primary Completion 2020-02-10 (Actual); Study Completion 2020-02-10 (Actual)

PRIMARY OUTCOMES:
Enrollment of eligible participants (accrual) | Up to 30 days post the end of the six-week program
  Feasibility will be assessed through enrollment of >= 60% of eligible participants (accrual) and completion of at least 5 out of 6 sessions for >= 80% of participants (adherence/engagement).
Completion of sessions (adherence/engagement) | Up to 30 days post the end of the six-week program
  Feasibility will be assessed through enrollment of >= 60% of eligible participants (accrual) and completion of at least 5 out of 6 sessions for >= 80% of participants (adherence/engagement).

SECONDARY OUTCOMES:
Change in Functional Assessment of Cancer Therapy-Cognition scores | Baseline up to 30 days post the end of the six-week program
  Functional Assessment of Cancer Therapy-Cognitive Function (version 3) (assesses cognitive functioning) The four subscales and associated ranges are as follows: Perceived Cognitive Impairments (range 0-72), Impact of Perceived Cognitive Impairments on Quality of Life (range 0-16), Comments from Others (range 0-16) and Perceived Cognitive Abilities (range 0-28).
  The higher the score, the better the outcome. There is no total score on this measure.
Change in Patient Reported Outcomes Measurement Information System (PROMIS) scores | Baseline up to 30 days post the end of the six-week program
  Will be used to characterize the change of the study population and evaluate patterns suggesting potential intervention efficacy on outcomes.
  Patient Reported Outcomes Measurement Information System: Cognitive Function- General Concerns version 1.0 and Cognitive Function-Abilities version 1.0 subscales (assess cognitive functioning).For each of these scales the raw score range is 8-40. These scores are then converted to T-scores (Mean = 50, SD = 10).For each of these scales the raw score range is 8-40. These scores are then converted to T-scores (Mean = 50, SD = 10).
  Subscales are not combined for these scales
Change in Global Self-Report of Cognition scores | Baseline up to 30 days post the end of the six-week program
  Will use two additional questions in an attempt to capture patient's perception of pre-treatment and current cognitive function and memory. These questions will be scored on a Likert scale (0= best memory possible, 10= worst memory possible) and will be provided to patients at the first and last session. Will be used to characterize the change of the study population and evaluate patterns suggesting potential intervention efficacy on outcomes.
Change in PROMIS-29 items (29) scores | Baseline up to 30 days post the end of the six-week program
  Each domain is scored separately. Will be used to characterize the change of the study population and evaluate patterns suggesting potential intervention efficacy on outcomes.
  Patient Reported Outcomes Measurement Information System-29 version 2.0 (assesses symptoms of depression, anxiety, physical function, pain interference, pain intensity, fatigue, sleep disturbance, and ability to participate in social and activities.
  Raw scores range from 4-20 for each subscale listed above except pain intensity which is a single item ranging from 0-10. The raw scores are then converted into T-scores (Mean = 50, SD = 10).
  For physical function, two sleep items and social activities subscales a higher T-score represents higher functioning. For anxiety, depression, fatigue, the other two sleep items and pain interference a higher T-score represents worse functioning.
  The subscales are not combined on this measure
Satisfaction Survey scores | Up to 30 days post the end of the six-week program
  Will use a survey to assess satisfaction with the class content and delivery. Will be used to characterize the change of the study population and evaluate patterns suggesting potential intervention efficacy on outcomes.
  Emerging From the Haze Course Survey (assesses satisfaction with the course and content).
  Total scores from responses range from 0-56. Higher values represent more satisfaction with the program. The scores are not combined for this survey.

CONTACTS AND LOCATIONS:
Overall Officials: Natalie Kelly, PhD, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States